CLINICAL TRIAL: NCT04233762
Title: The Effect of Sex Hormone Levels During the Menstrual Cycle on Capsaicin Evoked Cough
Brief Title: Effect of Sex Hormone During the Menstrual Cycle on Capsaicin Evoked Cough Responses
Acronym: CASH
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: McMaster-CASH
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Female Natural Cycle Group: Females with regular natural menstrual cycle.
- Female Oral Contraceptive Pill Group: Females taking the combined oral contraceptive pill.
- Male Group: Males with no history of anabolic steroid use.

SUMMARY:
The study aim is to investigate if changes in sex hormones during the menstrual cycle affects cough sensitivity in females and males with mild allergic asthma. Female subjects will be grouped according to natural cycle, or taking oral contraceptives. Male subjects will act as the control group.

DETAILED DESCRIPTION:
The study will have a total of 3 visits separated by at least 24 hours. Screening Period (Visits 1) - For All Subjects. Eligible subjects will be identified during the initial screening procedures with measures of spirometry, hyperresponsiveness to methacholine, complete history, physical examination, allergen skin test, and capsaicin cough challenge. For female subjects, this visit will occur during Day 1-5 (follicular phase) of the menstrual cycle. Subjects meeting the eligibility criteria will be randomized to Sequence A or Sequence B.

Sequence A will require Visit 2 to occur during menstrual cycle days 1-5 (follicular phase) and Visit 3 to occur during menstrual cycle days 21 - 25 (luteal phase).

Sequence B will require Visit 2 to occur during menstrual cycle days 21-25 (luteal phase) and Visit 3 to occur during menstrual cycle days 1 - 5 (follicular phase).

During Visit 2 and 3 subjects will undergo measures of spirometry, hyperresponsiveness to methacholine, capsaicin cough challenge, allergen skin test, sputum and blood collection.

Visit Windows Each visit must be separated by a minimum of 24 hours. Study visits can be performed in the morning or afternoon, however for each subject the timing should be consistent with Visit 1 at the same time of day ± 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be aged between 18 to 35 years
2. Have a diagnosis of atopic asthma (based on at least one positive skin prick test and methacholine PC20 ≤16 mg/ml)
3. FEV1 ≥ 70% of predicted
4. Demonstrate a cough response to capsaicin with a minimum of 3 coughs during the screening capsaicin challenge

Exclusion Criteria:

1. Subjects who are in a pollen season that affects their asthma
2. Subjects who report allergies to capsaicin or bronchoconstrict at the end of the full dose capsaicin cough challenge and require short acting bronchodilator therapy (assess after visit 1)
3. Subjects who do not display evidence of airway hyper-responsiveness (methacholine PC20>16mg/ml) (assess after visit 1)
4. Symptoms of upper respiratory tract infection in the last 1 month which have not resolved.
5. Lower respiratory tract infection or pneumonia in the last 6 weeks.
6. Current smoker or ex-smoker with ≥10 pack year smoking history and abstinence of ≤6 months
7. Asthma exacerbation in the previous month requiring a start of inhaled or oral corticosteroids.
8. Any asthma medication with the exception of infrequent (less than twice weekly) short-acting β2-agonist.
9. Subjects who have changed asthma medication within the past 4 weeks prior to screening
10. A previous asthma exacerbation requiring Intensive Care Unit admission.
11. Significant other primary pulmonary disorders in particularly; pulmonary embolism, pulmonary hypertension, interstitial lung disease, lung cancer, cystic fibrosis, emphysema or bronchiectasis.
12. Pregnancy or breast-feeding
13. Use of ACE inhibitors
14. Any centrally acting medication (opioids, gapapentin, pregabalin, amitriptyline) which in the view of the investigator could alter the sensitivity of the cough reflex
15. History of psychiatric illness, drug or alcohol abuse which may interfere in the participation of the trial.
16. History of current or previous anabolic steroid use in men.
17. For the natural cycle group, the female patients must have regular (24 to 35 day) natural cycles and no oral contraceptive use for ≥6 months
18. For female's taking the oral contraceptive pill they must be taking this ≥6 months
19. Use of B-blockers
20. Patients with clinically significant cardiovascular disease
21. Patients with known allergy to any of the study medications or excipients
22. Patients with a known potentially life threatening allergy (e.g. food allergy, stinging insect allergy), history of anaphylaxis, mastocytosis, angioedema

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mild atopic asthmatics
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Emax | One visit during day 1 to day 5 of the menstrual cycle, compared to one visit during day 21 to 25 of the menstrual cycle
  The maximum number of capsaicin evoked coughs

SECONDARY OUTCOMES:
ED 50 | One visit during day 1 to day 5 of the menstrual cycle, compared to one visit during day 21 to 25 of the menstrual cycle
  The dose of capsaicin that evokes at least half the maximum number of coughs(ED50) in days 1 -5 and 21 - 25 of the natural cycle, and between the natural cycle, male subjects and female subjects taking the oral contraceptive pill
Dose response Curve | One visit during day 1 to day 5 of the menstrual cycle, compared to one visit during day 21 to 25 of the menstrual cycle
  Changes in the capsaicin full dose response curves
C2 and C5 | One visit during day 1 to day 5 of the menstrual cycle, compared to one visit during day 21 to 25 of the menstrual cycle
  Changes in the dose of capsaicin causing 2 coughs (C2) and 5 coughs (C5)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — Professor Department of Medicine
Locations (1):
- McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No